CLINICAL TRIAL: NCT00001699
Title: A Pilot Study of Adherence to Oral Medication and Health Beliefs of Adolescents With HIV and Their Mothers
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 980121; 98-C-0121
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-06

CONDITIONS: Acquired Immunodeficiency Syndrome; HIV Infections
Keywords: AIDS; Compliance; HIV; Medication; Perceived Threat; Teenagers
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections; Patient Compliance

SUMMARY:
The proposed study has two specific aims 1) to gather data about treatment adherence levels among adolescents (11-21 years) with HIV and 2) to obtain information about the adolescents and mothers' health beliefs and examine their relationship to the adolescents' adherence levels. This pilot study is designed to gather preliminary data about the feasibility of using several new measures with this population. To achieve these aims, a convenience sample of approximately 45 adolescents with HIV will re recruited. The adolescents and their mothers will complete a brief questionnaire about their health beliefs. A 24-hour recall interview format will be used to assess the adolescents' treatment adherence to prescribed oral medication. The adolescent will complete recall interviews on three random days over a two week period. Data analysis will be primarily descriptive, but will be used to generate more specific hypotheses for future research studies. The long-term goal of this research is to better identify adolescents with HIV at risk for non-adherence and design empirically derived interventions to improve their adherence levels. The health beliefs measure may also be useful in identifying irrational beliefs about the illness or treatment that can then be targeted for cognitive restructing in psychological interventions.

DETAILED DESCRIPTION:
The proposed study has two specific aims 1) to gather data about treatment adherence levels among adolescents (11-21 years) with HIV and 2) to obtain information about the adolescents and mothers' health beliefs and examine their relationship to the adolescents' adherence levels. This pilot study is designed to gather preliminary data about the feasibility of using several new measures with this population. To achieve these aims, a convenience sample of approximately 45 adolescents with HIV will be recruited. The adolescents and their mothers will complete a brief questionnaire about their health beliefs. A 24-hour recall interview format will be used to assess the adolescents' treatment adherence to prescribed oral medication. The adolescent will complete recall interviews on three random days over a two week period. Data analysis will be primarily descriptive, but will be used to generate more specific hypotheses for future research studies. The long-term goal of this research is to better identify adolescents with HIV at risk for non-adherence and design empirically derived interventions to improve their adherence levels. The health beliefs measure may also be useful in identifying irrational beliefs about the illness or treatment that can then be targeted for cognitive restructing in psychological interventions.

ELIGIBILITY:
Subjects must be between the ages of 11 and 21 years.

Subjects must be diagnosed with HIV for at least one year (to ensure sufficient opportunity to experience living with a chronic condition such that adherence level is unlikely to be the result of skill or knowledge deficits).

Subjects must be prescribed oral medications (e.g., pills, liquids, inhaler) to be taken on a daily basis.

Subjects must be living with same female caregiver for at least one year.

Subjects must have a telephone number where he/she can be contacted during the two weeks after recruitment.

The adolescent and mother must be able to provide informed consent.

Adolescents must not have mental retardation or developmental delay that would prevent the adolescent from reading and comprehending the questionnaire.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45
Dates: Start 1998-06; Study Completion 2000-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Freund A, Johnson SB, Silverstein J, Thomas J. Assessing daily management of childhood diabetes using 24-hour recall interviews: reliability and stability. Health Psychol. 1991;10(3):200-8. doi: 10.1037//0278-6133.10.3.200. PMID 1879392
- [Background] Tamaroff MH, Festa RS, Adesman AR, Walco GA. Therapeutic adherence to oral medication regimens by adolescents with cancer. II. Clinical and psychologic correlates. J Pediatr. 1992 May;120(5):812-7. doi: 10.1016/s0022-3476(05)80257-4. PMID 1578322
- [Background] Becker MH, Maiman LA. Sociobehavioral determinants of compliance with health and medical care recommendations. Med Care. 1975 Jan;13(1):10-24. doi: 10.1097/00005650-197501000-00002. PMID 1089182